CLINICAL TRIAL: NCT02407509
Title: A Phase I Trial of VS-6766 (RO5126766) (a Dual RAF/MEK Inhibitor) Exploring Intermittent, Oral Dosing Regimens in Patients With Solid Tumours or Multiple Myeloma, With an Expansion to Explore Intermittent Dosing in Combination With Everolimus
Brief Title: Phase I Trial of VS-6766 Alone and in Combination With Everolimus
Acronym: RAF/MEK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Chugai Pharmaceutical (Industry); Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR3808; 2012-001040-22 (EudraCT Number)
Record Dates: First submitted 2015-02-09; First posted 2015-04-03 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumours; Multiple Myeloma; Lung Cancer; Ovarian Cancer
MeSH Terms: conditions — Multiple Myeloma; Lung Neoplasms; Ovarian Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part I - Twice weekly (COMPLETED) (Experimental): VS-6766 will be administered twice weekly in 4 week cycles in patients with solid tumours.
  Interventions: Drug: VS-6766
- Part I - Three times weekly (COMPLETED) (Experimental): VS-6766 will be administered three times weekly in 4 week cycles in patients with solid tumours.
  Interventions: Drug: VS-6766
- Part IIA (COMPLETED) (Experimental): VS-6766 will be administered twice weekly in 4 week cycles in patients with solid tumours with a mutation in the RAS-RAF-MEK pathway.
  Interventions: Drug: VS-6766
- Part IIB (CLOSED) (Experimental): VS-6766 will be administered twice weekly in 4 week cycles in patients with multiple myeloma with a mutation in KRAS, NRAS or BRAF. In order to accommodate steroid use for patients with multiple myeloma, patients will be administered for 3 weeks followed by a week interruption.
  Interventions: Drug: VS-6766
- Part IIC (COMPLETED) (Experimental): VS-6766 will be administered twice weekly in 4 week cycles in patients with solid tumours with a mutation in the RAS-RAF-MEK pathway. Upon occurrence of specified G2 toxicity, dosing intensity will be reduced to 3 weeks followed by a week interruption in a 4 week cycle.
  Interventions: Drug: VS-6766
- Part IID - Once weekly dose confirmation (COMPLETED) (Experimental): VS-6766 and everolimus will be administered once weekly in 4 week cycles in patients with solid tumours with a mutation in the RAS-RAF-MEK pathway. All patients will dose for 3 weeks followed by a week interruption in a 4 week cycle.
  Interventions: Drug: VS-6766; Drug: Everolimus
- Part IID - Twice weekly dose confirmation (COMPLETED) (Experimental): VS-6766 and everolimus will be administered twice weekly in 4 week cycles in patients with solid tumours with a mutation in the RAS-RAF-MEK pathway. All patients will dose for 3 weeks followed by a week interruption in a 4 week cycle.
  Interventions: Drug: VS-6766; Drug: Everolimus
- Part IID - Dose expansion (Experimental): VS-6766 and everolimus will be administered twice weekly in 4 week cycles in patients with KRAS-mutant lung cancer. All patients will dose for 3 weeks followed by a week interruption in a 4 week cycle.
  Interventions: Drug: VS-6766; Drug: Everolimus
- Part IIE- Biopsy Cohort (Experimental): VS-6766 and everolimus will be administered twice weekly in 4 week cycles in patients with documented RAS or RAF mutant solid tumours All patients will dose for 3 weeks followed by a week interruption in a 4 week cycle.
  Interventions: Drug: VS-6766; Drug: Everolimus
- Part IIF- LGSOC Cohort (Experimental): VS-6766 and everolimus will be administered twice weekly in 4 week cycles in patients with LGSOC who have previously been treated with the combination of VS-6766 and defactinib within 24 months of trial entry. Additionally, all patients must have displayed anti-tumour activity on the VS-6766 and defactinib combination, defined as follows:
  • Experienced a response - confirmed partial response (PR) or complete response (CR) - according to RECIST 1.1.
  Or
  • Experienced stable disease (SD) according to RECIST 1.1 (Appendix 3) AND patient received VS-6766 and defactinib treatment for a minimum of 12 months.
  All patients will dose for 3 weeks followed by a week interruption in a 4 week cycle.
  Interventions: Drug: VS-6766; Drug: Everolimus

INTERVENTIONS:
Drug: VS-6766
Drug: Everolimus
  Arms: Part IID - Dose expansion; Part IID - Once weekly dose confirmation (COMPLETED); Part IID - Twice weekly dose confirmation (COMPLETED); Part IIE- Biopsy Cohort; Part IIF- LGSOC Cohort

SUMMARY:
In Part I of the study VS-6766 will be given twice weekly or three times per week in treatment cycles of 4 weeks to investigate a safe and tolerable dose of the drug.

Once the optimal dosing schedule is defined, the following patients with BRAF, KRAS and/or NRAS mutations will be enrolled: 26 patients with solid tumours (Parts IIA & IIC) and 10 patients with Multiple Myeloma (Part IIB).

Up to 44 patients with solid tumours containing BRAF, KRAS and/or NRAS mutations will take VS-6766 in combination with everolimus (Part IID). Of these, 20 patients will comprise the Part IID dose expansion and will all have KRAS-mutant lung cancer.

DETAILED DESCRIPTION:
This is a two centre Phase I trial evaluating two intermittent dosing schedules of VS-6766 alone and then in combination with everolimus.

Part I (COMPLETED): Patients will be given VS-6766 (4mg) twice weekly or three times per week in treatment cycles of 4 weeks to investigate a safe and tolerable dose of the drug. Up to six patients will be enrolled to each dosing schedule and once they have completed 1 cycle of treatment the Safety Review Committee (SRC) will review their safety data, PK and PD data and define the optimal schedule to be taken forward into Part II.

On the basis of the previous Phase I trial, dose limiting toxicities (DLTs) are not expected at a dose of 4 mg but in the event of ≥ 2 DLT's occurring in (a) the 2 x weekly arm, then no further patients will recruited into that arm and the schedule will not be taken forward to Part II, or (b) the 3 x weekly arm, a single dose reduction to 3.2mg on the same dosing schedule will be implemented and 6 patients enrolled at the reduced dose. If 4 mg given 3 x weekly is considered non-tolerable, then the SRC may decide to enrol patients to the 3.2 mg dose level in the absence of dose limiting toxicity.

* If both the 2 x weekly (Mon & Thurs / Tues & Fri) and 3 x weekly (Mon, Wed & Fri) schedule are tolerated at 4 mg i.e. < 2 DLT's out of a 6 patients in each schedule, then the 3 x weekly schedule will be selected.
* If the 3 x weekly schedule requires a dose reduction to 3.2 mg and the 2 x weekly schedule is tolerated at 4 mg, then PD data will be evaluated relative to AUC to aid the selection.
* If ≥2 DLT's occur out of 6 patients in both schedules (despite the 3 x weekly arm being dose reduced), Part II will not be initiated and the study will be terminated.

Selection of the optimum schedule from Part I will be made by the Safety Review Committee and will be the schedule that delivers the highest, tolerable, cumulative weekly dose.

Part II: Once the optimal dosing schedule has been established in Part I, the following groups of patients will be enrolled:

Part IIA (COMPLETED) - 20 patients with documented RAS-RAF-MEK pathway mutant solid tumours (including KRAS, NRAS or BRAF).

Part IIB (CLOSED) - 10 patients with documented KRAS, NRAS or BRAF multiple myeloma.

NB: In order to accommodate steroid use for patients with multiple myeloma, the optimal dosing schedule as determined in Part I will be administered for 3 weeks followed by a week interruption.

Part IIC (COMPLETED) - An additional 6 patients with RAS-RAF-MEK pathway mutant solid tumours (including but not exclusive to KRAS, NRAS or BRAF) will be enrolled at the MTD determined in Part I however, upon occurrence of Grade 2 drug-related skin rash, CPK elevation or diarrhoea the dosing intensity will be reduced to 3 weeks followed by a week interruption. Of the six patients in Part IIC, at least three patients should have KRAS mutant lung cancer.

Part IID - a maximum of 44 patients with documented RAS-RAF-MEK pathway mutant solid tumours (including KRAS, NRAS and/or BRAF) will be administered with the combination of VS-6766 and everolimus for 3 weeks followed by a week interruption. Part IID will be split into two arms, dose confirmation and dose expansion:

* Part IID dose confirmation (COMPLETED) - Up to 24 patients will be treated at Schedule A (once-weekly dosing) or Schedule B (twice-weekly dosing). Each dose comprises 4mg VS-6766 + 5mg everolimus in combination. If Schedule A is tolerable, patients will be dosed at Schedule B. Should either of these schedules not be tolerable, the dose of VS-6766 can be reduced to 3.2mg.
* Part IID dose expansion (COMPLETED)- 20 patients will be treated at the optimal dosing schedule identified in Part IID dose confirmation. All patients will have KRAS-mutant lung cancer.
* Part IIE Biopsy Cohort - 6 patients will be treated at the optimal dosing schedule identified in Part IID dose expansion. Pharmacodynamic studies in pre- and post-treatment paired tumour biopsy samples will be investigated in this cohort, in addition to the plasma concentration of VS-6766 and everolimus at the time of on-treatment biopsies through pharmacokinetic analysis. Biopsies and blood draws for pharmacodynamic and pharmacokinetic assays will be mandatory.
* Part IIF LGSOC Cohort - 10 patients with LGSOC will be treated with the optimal dosing schedule identified in Part IID dose expansion. All patients in Part IIF will have been previously been treated with the combination of VS-6766 and defactinib within 24 months of trial entry.

ELIGIBILITY:
INCLUSION CRITERIA:

1. 18 years or over
2. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
3. Histologically or cytologically proven solid tumours or Multiple Myeloma refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient
4. Life expectancy of at least 12 weeks
5. World Health Organisation (WHO) performance status of 0 or 1
6. Measurable and/or evaluable disease according to RECIST 1.1 for patients with solid tumours or according to IMWG for multiple myeloma patients.
7. Haematological and biochemical indices within the ranges shown in the protocol. These measurements must be performed within two weeks (Day -14 to Day 1) before the patient is entered into the trial.

   ADDITIONAL INCLUSION CRITERIA FOR Part II:
8. Documented presence of RAS-RAF-MEK pathway mutations including BRAF, KRAS and NRAS. In Part IIC at least three patients should have KRAS mutant lung cancer. In Part IID expansion, all 20 patients should have KRAS mutant lung cancer.
9. Patients with multiple myeloma refractory to conventional treatment. Haematological indices as in section 4.1.1 above except ANC ≥ 1.0 x 10^9/L, platelet count ≥ 50 x 10^9/L and serum creatinine ≤ 1.5 x (ULN). Patients can be deemed as eligible based on serum creatinine alone if creatinine clearance/isotope clearance is deranged.
10. Archival tumour sections available for patients with solid tumours, or diagnostic bone marrow samples available for patients with multiple myeloma.

111. For patients with solid tumours only: presence of at least one measurable disease lesion according to RECIST 1.1.

Additional inclusion criteria for Part IIA, Part IIB, Part IIC, Part IID and Part IIE:

Documented presence of RAS-RAF-MEK pathway mutations including BRAF, KRAS and NRAS. In Part IIC at least three patients should have KRAS mutant lung cancer. In Part IID expansion, all 20 patients should have KRAS mutant lung cancer. In Part IIE, all 6 evaluable patients should have any RAS or RAF mutant solid tumours.

Additional inclusion criteria for Part IIE:

Patients must have disease that is amenable to biopsy and must be willing to undergo tumour biopsies (collected pre- and post-treatment). Patients must be willing to have blood draws for PK analysis (collected pre- and post-treatment).

Additional inclusion criteria for Part IIF:

Patients must have low-grade serous ovarian cancer (LGSOC) which has previously displayed anti-tumour activity on the combination treatment of VS-6766 and defactinib, where anti-tumour activity is defined as one of the following:

• A best response of confirmed complete response (CR) or partial response (PR), according to RECIST 1.1 (Appendix 3).

OR

• A best response of stable disease (SD), according to RECIST 1.1 (Appendix 3), AND received VS-6766 and defactinib combination treatment for a minimum of 12 months.

Patients must have received the combination treatment of VS-6766 and defactinib within 24 months of the first dose of either study drug.

EXCLUSION CRITERIA:

1. Prior chemotherapy, radiotherapy (other than a short cycle of palliative radiotherapy for bone pain), or immunotherapy within 28 days of first receipt of study drug (within 6 weeks for nitrosoureas and mitomycin C), with the exception of Dexamethasone for patients with multiple myeloma. Hormone therapy within 14 days of first receipt of study drug, with exception of prostate cancer if indicated. In patients with brain metastases, previous radiotherapy should have finished at least 28 days prior and limited steroid management is required. Steroid management should not exceed 4mg dexamethasone, or equivalent, per day.
2. Ongoing toxic manifestations of previous treatments except Grade 1 toxicities which in the opinion of the Investigator should not exclude the patient.
3. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
4. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
5. Major thoracic or abdominal surgery from which the patient has not yet recovered.
6. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
7. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
8. Patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease.
9. History of any bowel disease including abdominal fistula, gastro-intestinal perforation, and diverticulitis.
10. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA] - refer to Appendix 5), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease.
11. Concurrent ocular disorders:

    1. Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes, uncontrolled hyperlipidemia, uncontrolled hypercholesterolemia, hyperviscosity syndromes, medically significant history of vasculitis, inflammatory, atherosclerotic or thrombophilic conditions and coagulopathy.
    2. Patient with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
    3. Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions
12. Patients exposed to CYP3A4 inhibitors within 7 days prior to the first dose.
13. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of VS-6766 and/or everolimus. Participation in an observational trial would be acceptable.
14. Symptoms of COVID-19 and/or documented current COVID-19 infection (the patient can be reassessed for eligibility following a full recovery and negative COVID-19 test)
15. Any other condition which in the Investigator's opinion would not make the patient a good candidate for a clinical trial with VS-6766 e.g. hypersensitivity to VS-6766.

Part IID, Part IIE and Part IIF specific exclusions:

1. Has received a live vaccine within 30 days of planned start of study therapy. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
2. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   Diagnosis of diabetes mellitus types I or II (irrespective of management). Glycosylated haemoglobin (HbA1C) ≥7.0% at screening Fasting Plasma Glucose ≥ 8.3mmol/L at screening. Fasting is defined as no caloric intake for at least 8 hours.
3. Any other condition which in the Investigator's opinion would not make the patient a good candidate for a clinical trial with Everolimus. Examples of which include: hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption; hypersensitivity to Everolimus, to other rapamycin derivatives or to any of the excipients; pre-existing infections.

   Additional exclusion criteria for Part IIF:
4. Patients that have previously discontinued treatment of VS-6766 and/or defactinib for reasons of toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2013-06-17 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Recommend a phase II dose and dosing schedule for VS-6766, as a single agent and also in combination with everolimus. | In the first cycle of treatment (28-35 days).
  Determining the schedule at which no more than one patient out of six patients experience a highly probable or probable drug-related dose limiting toxicity.
Assess the safety and toxicity profile of each schedule of administration of VS-6766 both as a single agent and in combination with everolimus. | Throughout time on trial per patient, estimated to be 6 months.
  Determining causality of each adverse event to VS-6766 and everolimus, grading severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

SECONDARY OUTCOMES:
Determining the pharmacokinetic profile of VS-6766 - Cmax | In the first cycle of treatment (28-35 days).
  Determining Peak Plasma Concentration (Cmax) of VS-6766 given via intermittent dosing schedules in selected patients.
Determining the pharmacokinetic profile of VS-6766 - AUC | In the first cycle of treatment (28-35 days).
  Determining the Area under the plasma concentration versus time curve (AUC) of VS-6766 given via intermittent dosing schedules in selected patients.
Determining the pharmacokinetic profile of VS-6766 - T½ | In the first cycle of treatment (28-35 days).
  Determining the half-life (T½) of VS-6766 given via intermittent dosing schedules in selected patients.
Determining the pharmacokinetic profile of VS-6766 - Accumulation index | In the first cycle of treatment (28-35 days).
  Determining the accumulation index of VS-6766 given via intermittent dosing schedules in selected patients.
Determining the pharmacodynamic profile of VS-6766 | In the first cycle of treatment (28-35 days).
  Quantifying pERK levels in PBMCs in selected patients.
Determining anti-tumour activity of VS-6766, as a single agent and also in combination with everolimus. | Throughout time on trial per patient, estimated to be 6 months.
  Anti-tumour activity is any response (stable disease, partial response or complete response) in any of the patients as determined by the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.

OTHER OUTCOMES:
Pharmacodynamic studies in optional pre- and post-treatment paired tumour biopsy samples in selected patients. | In the first cycle of treatment (28-35 days).
  Quantifying downstream activation of signal transduction and cell death.
Exploratory Functional Imaging Studies | Throughout time on trial per patient, estimated to be 6 months.
  Review of diffusion-weighted (DW)-MRI, 1H-MRS (Magnetic Resonance Spectroscopy) and 18F-choline positron emission tomography (PET) imaging scans for exploration of predictive imaging biomarkers of response in selected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, MBBS, PhD, Principal Investigator — The Institute of Cancer Research, Royal Marsden NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Guy's and St Thomas' Hospital, London
  - Gynaecological Unit - Royal Marsden NHS Foundation Trust, London

REFERENCES:
- [Derived] Guo C, Chenard-Poirier M, Roda D, de Miguel M, Harris SJ, Candilejo IM, Sriskandarajah P, Xu W, Scaranti M, Constantinidou A, King J, Parmar M, Turner AJ, Carreira S, Riisnaes R, Finneran L, Hall E, Ishikawa Y, Nakai K, Tunariu N, Basu B, Kaiser M, Lopez JS, Minchom A, de Bono JS, Banerji U. Intermittent schedules of the oral RAF-MEK inhibitor CH5126766/VS-6766 in patients with RAS/RAF-mutant solid tumours and multiple myeloma: a single-centre, open-label, phase 1 dose-escalation and basket dose-expansion study. Lancet Oncol. 2020 Nov;21(11):1478-1488. doi: 10.1016/S1470-2045(20)30464-2. Epub 2020 Oct 28. PMID 33128873